CLINICAL TRIAL: NCT06022939
Title: A Phase III, Randomized Study of Daratumumab, Cyclophosphamide, Bortezomib and Dexamethasone (Dara-VCD) Induction Followed by Autologous Stem Cell Transplant or Dara-VCD Consolidation and Daratumumab Maintenance in Patients With Newly Diagnosed AL Amyloidosis
Brief Title: Comparing Dara-VCD Chemotherapy Plus Stem Cell Transplant to Dara-VCD Chemotherapy Alone for People Who Have Newly Diagnosed AL Amyloidosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: S2213; NCI-2023-04234 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2213 (Other: SWOG); S2213 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2023-08-11; First posted 2023-09-05 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: AL Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — Stem Cell Transplantation; Biopsy; Specimen Handling; Bortezomib; Cyclophosphamide; daratumumab; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Magnetic Resonance Spectroscopy; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Consolidation Arm I (Chemotherapy) (Active Comparator): Patients receive daratumumab and hyaluronidase-fihj SC over 3-5 minutes on days 1 and 15 as well as bortezomib SC over 3-5 minutes, cyclophosphamide PO or IV, and dexamethasone PO or IV on days 1, 8, 15 and 22 of each cycle. Cycles repeat every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography at screening and at progression. Patients undergo bone marrow aspiration and biopsy within14-28 days post consolidation treatment and at progression. Patients undergo blood and urine sample collection at screening, at the start of each cycle, and the end of treatment and during follow up or at progression.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Bortezomib; Drug: Cyclophosphamide; Drug: Daratumumab and Hyaluronidase-fihj; Drug: Dexamethasone; Procedure: Echocardiography; Other: Survey Administration
- Consolidation Arm II (Chemotherapy, ASCT) (Experimental): Patients undergo collection of peripheral blood stem cells. Patients receive melphalan IV for 1 cycle and then 2 days later receive the stem cell transplant IV in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography at screening and at progression. Patients undergo bone marrow aspiration and biopsy within 60-90 days post initiation of stem cell transplant. Patients undergo blood and urine sample collection at screening, during treatment, and the end of treatment and during follow up or at progression.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Echocardiography; Drug: Melphalan; Procedure: Stem Cell Isolation; Other: Survey Administration
- Induction (Chemotherapy) (Experimental): Patients receive daratumumab and hyaluronidase-fihj SC over 3-5 minutes on days 1, 8, 15 and 22 for 2 cycles and then days 1 and 15 for cycle 3. Patients receive bortezomib SC over 3-5 minutes, cyclophosphamide PO or IV, and dexamethasone PO or IV on days 1, 8, 15 and 22 of each cycle. Cycles repeat every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT, MRI or PET-CT and fat pad aspiration at screening. Patients undergo echocardiography at screening, the completion of induction, and at progression. Patients undergo bone marrow aspiration and biopsy at screening, post induction treatment and at progression. Patients undergo blood and urine sample collection at screening, at the start of each cycle, and the end of treatment and during follow up or at progression.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Bortezomib; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Daratumumab and Hyaluronidase-fihj; Drug: Dexamethasone; Procedure: Echocardiography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Survey Administration
- Maintenance (daratumumab and hyaluronidase-fihj) (Experimental): Patients receive maintenance daratumumab and hyaluronidase-fihj SC over 3-5 minutes on day 1 of each cycle. Cycles repeat every 28 days for up 18 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography at screening, 12 months post consolidation treatment and at progression. Patients undergo bone marrow aspiration and biopsy 12 months post consolidation treatment and at progression. Patients undergo blood and urine sample collection at screening, during treatment, 12 months post consolidation treatment and during follow up or at progression.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Daratumumab and Hyaluronidase-fihj; Procedure: Echocardiography; Other: Survey Administration

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Given IV
  Other Names: AHSCT; Autologous; Autologous Hematopoietic Cell Transplantation; Autologous Stem Cell Transplant; Autologous Stem Cell Transplantation; Stem Cell Transplantation, Autologous
  Arms: Consolidation Arm II (Chemotherapy, ASCT)
Procedure: Biopsy — Undergo fat pad biopsy
  Other Names: BIOPSY_TYPE; Bx
  Arms: Induction (Chemotherapy)
Procedure: Biospecimen Collection — Undergo blood and urine specimen collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Bortezomib — Given SC
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
  Arms: Consolidation Arm I (Chemotherapy); Induction (Chemotherapy)
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
  Arms: Induction (Chemotherapy)
Drug: Cyclophosphamide — Given PO or IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
  Arms: Consolidation Arm I (Chemotherapy); Induction (Chemotherapy)
Drug: Daratumumab and Hyaluronidase-fihj — Given SC
  Other Names: DARA Co-formulated with rHuPH20; DARA/rHuPH20; Daratumumab + rHuPH20; Daratumumab with rHuPH20; Daratumumab-rHuPH20; Daratumumab/Hyaluronidase-fihj; Daratumumab/rHuPH20 Co-formulation; Darzalex Faspro; Darzalex/rHuPH20; HuMax-CD38-rHuPH20; Recombinant Human Hyaluronidase Mixed with Daratumumab
  Arms: Consolidation Arm I (Chemotherapy); Induction (Chemotherapy); Maintenance (daratumumab and hyaluronidase-fihj)
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
  Arms: Consolidation Arm I (Chemotherapy); Induction (Chemotherapy)
Procedure: Echocardiography — Undergo echocardiography
  Other Names: EC
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
  Arms: Induction (Chemotherapy)
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
  Arms: Consolidation Arm II (Chemotherapy, ASCT)
Procedure: Positron Emission Tomography — Undergo PET-CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
  Arms: Induction (Chemotherapy)
Procedure: Stem Cell Isolation — Undergo stem cell collection
  Other Names: Isolation, Stem Cell; Stem Cell Collection; Stem Cell Recovery
  Arms: Consolidation Arm II (Chemotherapy, ASCT)
Other: Survey Administration — Ancillary study

SUMMARY:
This phase III trial compares the effect of adding a stem cell transplant with melphalan after completing chemotherapy with daratumumab, cyclophosphamide, bortezomib and dexamethasone (Dara-VCD) versus chemotherapy with Dara-VCD alone for treating patients with newly diagnosed amyloid light chain (AL) amyloidosis. Melphalan is a chemotherapy given prior to a stem cell transplant. Giving chemotherapy before a peripheral blood stem cell transplant helps kill cancer cells in the body and helps make room in the patient's bone marrow for new blood-forming cells (stem cells) to grow. The stem cells are then returned to the patients to replace the blood forming cells that were destroyed by the chemotherapy. Daratumumab is in a class of medications called monoclonal antibodies. It binds to a protein called CD38, which is found on some types of immune cells and cancer cells, including myeloma cells. Daratumumab may block CD38 and help the immune system kill cancer cells. Chemotherapy drugs, such as cyclophosphamide and bortezomib, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Dexamethasone is in a class of medications called corticosteroids. It is used to lower the body's immune response to help stop the growth of cancer cells. Giving a stem cell transplant with melphalan after Dara-VCD may kill more cancer cells in patients with newly diagnosed AL amyloidosis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare major organ deterioration progression-free survival between participants randomized to the autologous stem cell transplant (ASCT) and non-ASCT arms of this study.

SECONDARY OBJECTIVES:

I. To compare overall survival (OS) between participants randomized to the ASCT and non-ASCT arms of this study.

II. To compare rates of cardiac and renal organ responses between participants randomized to the ASCT and non-ASCT arms of this study.

III. To compare rates of cardiac and renal organ progression between participants randomized to the ASCT and non-ASCT arms of the study.

IV. To compare the frequency and severity of toxicities between participants randomized to the ASCT and non-ASCT arms of this study.

V. To compare minimal residual disease (MRD) negativity rates between participants randomized to the ASCT and non-ACST arms of this study.

ADDITIONAL OBJECTIVES:

I. To compare the best overall hematologic response rates between participants randomized to the ASCT and non-ASCT arms of this study.

II. To compare rates of hematologic complete response (CR) and very good partial response, following completion of consolidation therapy between participants randomized to the ASCT and non-ASCT arms of this study, post-consolidation.

III. To compare hematologic progression-free survival between participants randomized to the ASCT and non-ASCT arms of this study.

IV. To compare time to next treatment between participants randomized to the ASCT and non-ASCT arms of the study.

V. To evaluate utilization of delayed ASCT in participants randomized to the non-ASCT arm of the study.

TRANSLATIONAL MEDICINE PRIMARY OBJECTIVES:

I. To compare MRD negativity rates from bone marrow aspirates via next generation flow cytometry (NGF) between the ASCT and non-ASCT arms of this study post-consolidation.

II. To bank specimens for future use.

TRANSLATIONAL MEDICINE EXPLORATORY OBJECTIVES:

I. To evaluate MRD negativity rates at post-induction, and compare MRD negativity rates at 12 months post-consolidation from bone marrow aspirates via NGF between participants randomized to the ASCT and non-ASCT arms of this study.

II. To investigate the association of achieving MRD negativity at any point (post-induction, post-consolidation, or 12 months post-consolidation) via NGF from bone marrow aspirates with major organ deterioration-progression free survival (MOD-PFS).

III. To investigate the association of achieving sustained MRD negativity (MRD negative at two consecutive measurements -- post-induction, post-consolidation, and 12 months post-consolidation) via NGF from bone marrow aspirates with MOD-PFS.

QUALITY OF LIFE (QOL) PRIMARY OBJECTIVE:

I. To compare patient-reported physical function following consolidation treatment between participants randomized to the ASCT and non-ASCT arms using the Patient Reported Outcomes Measurement Information System (PROMIS)-29+2 Profile version (v) 2.1 physical function sub-scale.

QOL SECONDARY OBJECTIVES:

I. To compare patient-reported fatigue following consolidation treatment between participants randomized to the ASCT and non-ASCT arms using the PROMIS-29 fatigue subscale.

II. To compare longitudinal changes in physical function using the PROMS-29+2 between participants randomized to the ASCT and non-ASCT arms.

QOL EXPLORATORY OBJECTIVES:

I. To assess baseline symptom burden in AL amyloidosis patients prior to induction therapy using the PROMIS-29+2.

II. To compare mean scores of symptom scales using the PROMIS-29+2 following consolidation treatment, and at 6 months and 12 months from step 3 registration between treatment arms.

III. To compare mean scores of functional scales using the PROMIS-29+2, following consolidation treatment, and at 6 months and 12 months from step 3 registration between treatment arms.

IV. To explore whether longitudinal changes in symptoms, functioning, and overall heath related quality of life (HRQoL) as assessed by the PROMIS-29 +2 (version 2.1) differ according to treatment group and, separately, according to baseline cardiac or renal involvement using interaction tests between participants randomized to the ASCT and non-ASCT arms.

V. To compare health utility indices using the PROMIS preference score (PROPr) between patients randomized to the ASCT and non-ASCT arms.

PATIENT REPORTED OUTCOME (PRO)-COMMON TERMINOLOGY CRITERIA FOR ADVERSE EVENTS (CTCAE) PRIMARY OBJECTIVE:

I. To compare patient reported symptoms regarding treatment emergent adverse events of interest using the Patient Reported Outcome CTCAE (PRO-CTCAE) Measurement System between patients randomized to the ASCT and non-ASCT arms of this study.

OUTLINE:

INDUCTION: Patients receive daratumumab and hyaluronidase-fihj subcutaneously (SC) over 3-5 minutes on days 1, 8, 15 and 22 for 2 cycles and then days 1 and 15 for cycle 3. Patients receive bortezomib SC over 3-5 minutes, cyclophosphamide orally (PO) or intravenously (IV), and dexamethasone PO or IV on days 1, 8, 15 and 22 of each cycle. Cycles repeat every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT), magnetic resonance imaging (MRI) or positron emission tomography (PET)-CT and fat pad aspiration at screening. Patients undergo echocardiography at screening, the completion of induction, and at progression. Patients undergo bone marrow aspiration and biopsy at screening, post induction treatment and at progression. Patients undergo blood and urine sample collection at screening, at the start of each cycle, and the end of treatment and during follow up or at progression.

CONSOLIDATION: Patients who achieve an overall response of partial response or better after 3 cycles of Dara-VCD are randomized to 1 of 2 arms.

ARM I: Patients receive daratumumab and hyaluronidase-fihj SC over 3-5 minutes on days 1 and 15 as well as bortezomib SC over 3-5 minutes, cyclophosphamide PO or IV, and dexamethasone PO or IV on days 1, 8, 15 and 22 of each cycle. Cycles repeat every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography at screening and at progression. Patients undergo bone marrow aspiration and biopsy within14-28 days post consolidation treatment and at progression. Patients undergo blood and urine sample collection at screening, at the start of each cycle, and the end of treatment and during follow up or at progression.

ARM II: Patients undergo collection of peripheral blood stem cells. Patients receive melphalan IV for 1 cycle and then 2 days later receive the stem cell transplant IV in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography at screening and at progression. Patients undergo bone marrow aspiration and biopsy within 60-90 days post initiation of stem cell transplant. Patients undergo blood and urine sample collection at screening, during treatment, and the end of treatment and during follow up or at progression.

MAINTENANCE: Patients receive maintenance daratumumab and hyaluronidase-fihj SC over 3-5 minutes on day 1 of each cycle. Cycles repeat every 28 days for up 18 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography at screening, 12 months post consolidation treatment and at progression. Patients undergo bone marrow aspiration and biopsy 12 months post consolidation treatment and at progression. Patients undergo blood and urine sample collection at screening, during treatment, 12 months post consolidation treatment and during follow up or at progression.

After completion of study treatment, patients are followed up every 3 or 6 months up to 4 years after registration.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1: Participants must have systemic AL amyloidosis which is biopsy proven and includes histologically-confirmed by positive Congo red stain with green birefringence on polarized light microscopy, OR characteristic appearance by electron microscopy AND confirmatory AL amyloid typing (mass spectrometry-based proteomic analysis or immunofluorescence). If there is question regarding diagnosis, consult study chairs prior to registration
* STEP 1: Participants must have measurable disease within 28 days prior to treatment if initiated prior to registration or within 28 days of registration as defined by at least one of the following:

  * Positive monoclonal serum immunofixation electrophoresis
  * Positive monoclonal urine immunofixation electrophoresis
  * Monoclonal plasma cells in bone marrow In addition, participants must also have a difference between the involved and uninvolved free light chain (dFLC) >= 2 mg/dL
* STEP 1: Participants may receive up to one cycle (or 28 days) of therapy prior to enrollment. If a patient receives >= 75% of 1 cycle of protocol identical Dara-VCD, this will be considered 1 cycle of protocol induction. Any patient who receives less than 75% of 1 cycle of Dara-VCD or non-protocol therapy will still be eligible but will be treated per protocol. If protocol identical therapy is initiated prior to enrollment, this treatment is not continued but rather treatment is dictated per protocol
* STEP 1: Participants may be receiving chronic corticosteroids if they are being given for disorders other than AL amyloidosis or myeloma
* STEP 1: Participant must be >= 18 years old
* STEP 1: Participant must have Eastern Cooperative Oncology Group (ECOG) performance score (PS) of 0, 1, or 2 (PS = 3 may be allowed if secondary to neuropathy)
* STEP 1: Participant must have a complete medical history and physical exam within 28 DAYS prior to registration
* STEP 1: Participants must be willing to undergo high dose chemotherapy and autologous stem cell transplantation if they are randomized to the arm receiving high dose chemotherapy and autologous stem cell transplantation
* STEP 1: Participants must be eligible to receive high dose chemotherapy with melphalan at a dose of 200 mg/m^2 or 140 mg/m^2 (200 mg/m^2 is highly encouraged but not mandated). Transplant eligibility criteria are included in the general eligibility criteria listed below:

  * Participant must have a supine systolic blood pressure (BP) >= 90 mmHg (at registration step-1, this may by supported by midodrine
  * Participant must have non-severe cardiac AL (meeting all the below criteria) as defined by:

    * N-terminal proB-type natriuretic peptide (NT proBNP) < 5000 (if no NTproBNP, brain natriuretic peptide [BNP] must be available and < 400)
    * Troponin T (TnT) < 0.06. If not available, one of the following two criteria must be met:

      * High sensitivity troponin (hsTnT) T < 75 or troponin I < 0.1ng/dL
    * New York Heart Association (NYHA) I or II
    * Cardiac ejection fraction (EF) >= 40%
* STEP 1: Hemoglobin >= 8.0 g/dL (> 5 mmol/L); red blood cell transfusion allowed up to 7 day prior to registration (within 28 days prior to registration) (NOTE: Growth factor support granulocyte colony-stimulating factor [G-CSF] is permitted per institutional guidelines)
* STEP 1: Leukocytes >= 2 x 10^3/uL (within 28 days prior to registration) (NOTE: Growth factor support [G-CSF] is permitted per institutional guidelines)
* STEP 1: Absolute neutrophil count >= 1.0 x 10^3/uL (within 28 days prior to registration) (NOTE: Growth factor support [G-CSF] is permitted per institutional guidelines)
* STEP 1: Platelets >= 50 x 10^3/uL (within 28 days prior to registration) (NOTE: Growth factor support [G-CSF] is permitted per institutional guidelines)
* STEP 1: Total bilirubin =< 1.5 times the institutional upper limit of normal (ULN) unless history of Gilbert's disease. Participants with history of Gilbert's disease must have total bilirubin =< 5 x institutional ULN (within 28 days prior to registration)
* STEP 1: Direct bilirubin =< 2.0 mg/dL (within 28 days prior to registration)
* STEP 1: Aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) =< 3x upper limit of normal (ULN) (except if secondary to hepatic involvement) (within 28 days prior to registration)
* STEP 1: Alkaline phosphatase =< 750 U/L (except if secondary to hepatic involvement) (within 28 days prior to registration)
* STEP 1: Participants must have a serum creatinine =< the institutional (I)ULN OR measured OR calculated creatinine clearance >= 30 mL/min using the following Cockcroft-Gault formula. This specimen must have been drawn and processed within 28 days prior to registration
* STEP 1: If peripheral neuropathy is present at diagnosis, participants must be grade 2 (moderate symptoms; limiting instrumental activity of daily living [ADL]) or less
* STEP 1: Participants must have adequate cardiac function. Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants must be class 2 or better
* STEP 1: Participants must not be seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (i.e., subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR
* STEP 1: Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants currently being treated for HCV infection must have undetectable HCV viral load test on the most recent test results obtained within 6 months prior to registration, if indicated
* STEP 1: Participants must not have concurrent multiple myeloma as defined by the presence of lytic bone disease, plasmacytomas, >= 60% plasma cells in the bone marrow, or hypercalcemia. Participants will not be excluded solely based on the presence of plasma cells > 10% in the bone marrow unless the plasma cell percentage exceeds >60%
* STEP 1: Participants must not have known allergies to any of the study drugs
* STEP 1: Participants must not have had a major surgery within 14 days prior to registration and be fully recovered from surgery completed within 14 days prior to registration
* STEP 1: Participants must not have a known chronic obstructive pulmonary disease with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal
* STEP 1: Participants with known human immunodeficiency virus (HIV)-infection must be on effective anti-retroviral therapy at registration and have undetectable viral load test on the most recent test results obtained within 6 months prior to registration
* STEP 1: Participants must not have either moderate or severe persistent asthma within the past 2 years), or currently have uncontrolled asthma of any classification. (Note that subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed in the study)
* STEP 1: Participants must not have uncontrolled diabetes within 28 days prior to registration
* STEP 1: Participants must not have uncontrolled blood pressure and hypertension within 14 days prior to registration. Participants must have a supine systolic BP of >= 90 mmHg
* STEP 1: Participants must not have a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* STEP 1: Participants must not have received vaccination with live attenuated vaccines within 28 days prior to Registration to Step 1
* STEP 1: Participants must not have uncontrolled infection at the discretion of the enrolling physician and to be discussed with the study chair if the participant is on active anti-infectious therapy. Any patient on active anti-microbial therapy for chronic infectious issues should be discussed with the study chair prior to enrollment
* STEP 1: Participants must not be pregnant or nursing (nursing includes breast milk fed to an infant by any means, including from the breast, milk expressed by hand, or pumped). Individuals who are of reproductive potential must have agreed to use an effective contraceptive method with details provided as a part of the consent process. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen
* STEP 1: Participants must be offered the opportunity to participate in specimen banking. With participant consent, specimens must be collected and submitted via the Southwestern Oncology group (SWOG) Specimen Tracking System
* STEP 1: Participants must agree to have blood, bone marrow core biopsy and aspirate, and fat pad biopsy specimens submitted for minimal residual disease assessment and future exploratory studies
* STEP 1: Participants who can complete PRO, QOL, PRO-CTCAE questionnaires, etc. forms in English, Spanish and French must participate in the patient-reported outcomes and quality of life
* STEP 2: Participants must have met all eligibility criteria for Step-1 registration
* STEP 2: Participants must have achieved at least a partial response
* STEP 2: Participants must continue receiving at least one of study drugs (bortezomib, cyclophosphamide, or daratumumab and hyaluronidase-fihj) if another study drug (daratumumab and hyaluronidase-fihj, cyclophosphamide, or bortezomib) has been discontinued due to adverse events. Note: daratumumab and hyaluronidase-fihj cannot be permanently discontinued
* STEP 2: Participants must have completed induction therapy
* STEP 2: Participants must be registered to Step 2 within 42 days of cycle 3, day 28 of induction therapy
* STEP 2: Participants must plan to initiate their assigned consolidation therapy within 8 weeks after randomization
* STEP 2: Participants must not have experienced a MOD-PFS event
* STEP 2: Participants must have ECOG performance score (PS) of 0, 1, or 2 (PS = 3 may be allowed if secondary to neuropathy)
* STEP 2: Participant must have a complete medical history and physical exam within 28 days prior to registration
* STEP 2: Participants must be willing to undergo high dose chemotherapy and autologous stem cell transplantation if they are randomized to the arm receiving high dose chemotherapy and autologous stem cell transplantation
* STEP 2: Participants randomized to Arm 2 must be willing and able to return to a participating treatment center for their assigned treatment after transplant. Note that participants need not to have a direct relationship with the transplant center in order to register
* STEP 2: Participants must be eligible to receive high dose chemotherapy with melphalan at a dose of 200 mg/m^2 or 140 mg/m^2 (200 mg/m^2 is highly encouraged but not mandated). Transplant eligibility criteria are included in the general eligibility criteria listed below:

  * Patient must have a supine systolic BP >= 90 mmHg (at registration step-1, this may not by supported by midodrine)
  * Patient must have non-severe cardiac AL as defined by:

    * NT proBNP <5000 (if no NTproBNP, BNP must be available and < 400 pg/mL) (within 14 days prior to registration step-2)
    * TnT < 0.06. If not available, one of the following two criteria must be met (within 14 days prior to registration step-2)

      * hsTnT <75 or troponin I < 0.1ng/dL
    * NYHA I or II (within 14 days prior to registration step-2)
    * Cardiac EF >= 40% (within 14 days prior to registration step-2)
* STEP 2: Hemoglobin > 8.0 g/dL (> 5 mmol/L); red blood cell transfusion allowed up to 7 days prior to registration (within 28 days prior to registration) (NOTE: Growth factor support [G-CSF] is permitted per institutional guidelines)
* STEP 2: Leukocytes >= 2 x 10^3/uL (within 28 days prior to registration) (NOTE: Growth factor support [G-CSF] is permitted per institutional guidelines)
* STEP 2: Absolute neutrophil count >= 1.0 x 10^3/uL (within 28 days prior to registration) (NOTE: Growth factor support [G-CSF] is permitted per institutional guidelines)
* STEP 2: Platelets >= 50 x 10^3/uL (within 28 days prior to registration) (NOTE: Growth factor support [G-CSF] is permitted per institutional guidelines)
* STEP 2: Total bilirubin =< 1.5 times the institutional ULN unless history of Gilbert's disease. Participants with history of Gilbert's disease must have total bilirubin =< 5 x institutional ULN (within 28 days prior to registration)
* STEP 2: Direct bilirubin =< 2.0 mg/dL (except if secondary to hepatic involvement) (within 28 days prior to registration)
* STEP 2: AST/ALT =< 3x upper limit of normal (ULN) (except if secondary to hepatic involvement) (within 28 days prior to registration)
* STEP 2: Alkaline phosphatase =< 750 U/L (except if secondary to hepatic involvement) (within 28 days prior to registration)
* STEP 2: Participants must have a serum creatinine =< the IULN OR calculated creatinine clearance ≥ 30 mL/min using the following Cockcroft-Gault Formula. This specimen must have been drawn and processed within 28 days prior to registration
* STEP 2: Participants must not have uncontrolled infection at the discretion of the enrolling physician and to be discussed with the study chair if the participant is on active anti-infectious therapy. Any patient on active anti-microbial therapy for chronic infectious issues should be discussed with the study chair prior to enrollment
* STEP 2: Participants randomized to the ASCT arm must be able to have at least 2.0 x 10^6 CD34 cells/kg collected
* STEP 2: Participants who can complete PRO, QOL, PRO-CTCAE questionnaires, etc. forms in English, Spanish and French must participate in the patient-reported outcomes and quality of life
* STEP 3: Participants must have met all eligibility criteria for Step-1 and Step-2 registration
* STEP 3: Participants must not have had daratumumab and hyaluronidase-fihj permanently discontinued during induction or consolidation
* STEP 3: Participants must have completed induction and consolidation therapy
* STEP 3: Participants must be registered to Step 3 within the following time frames:

  * If randomized to Arm 1 Dara-VCD consolidation: within 28 days of completion of 3 cycles of consolidation therapy
  * If randomized to Arm 2 high dose chemotherapy and autologous stem cell transplantation: within 180 days following initiation of stem cell transplantation
* STEP 3: Participants must not have experienced a MOD-PFS event
* STEP 3: Participants must have ECOG performance score (PS) of 0, 1, or 2 (PS = 3 is allowed if secondary to neuropathy)
* STEP 3: Participants must have a complete medical history and physical exam within 28 DAYS prior to registration
* STEP 3: Hemoglobin > 8.0 g/dL (> 5 mmol/L); red blood cell transfusion allowed up to 7 days prior to registration (within 28 days prior to registration) (NOTE: Growth factor support [G-CSF] is permitted per institutional guidelines)
* STEP 3: Leukocytes >= 2 x 10^3/uL (within 28 days prior to registration) (NOTE: Growth factor support [G-CSF] is permitted per institutional guidelines)
* STEP 3: Absolute neutrophil count >= 1.0 x 10^3/uL (within 28 days prior to registration) (NOTE: Growth factor support [G-CSF] is permitted per institutional guidelines)
* STEP 3: Platelets >= 50 x 10^3/uL (within 28 days prior to registration) (NOTE: Growth factor support [G-CSF] is permitted per institutional guidelines)
* STEP 3: Total bilirubin =< 1.5 times the institutional upper limit of normal (ULN) unless history of Gilbert's disease. Participants with history of Gilbert's disease must have total bilirubin =< 5 x institutional ULN (within 28 days prior to registration)
* STEP 3: Direct bilirubin =< 2.0 mg/dL (within 28 days prior to registration)
* STEP 3: AST/ALT =< 3x upper limit of normal (ULN) (except if secondary to hepatic involvement) (within 28 days prior to registration)
* STEP 3: Alkaline phosphatase =< 750 U/L (except if secondary to hepatic involvement) (within 28 days prior to registration)
* STEP 3: Participants must not have uncontrolled infection at the discretion of the enrolling physician and to be discussed with the study chair if the participant is on active anti-infectious therapy. Any patient on active anti-microbial therapy for chronic infectious issues should be discussed with the study chair prior to enrollment
* Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines.

For participants with impaired decision-making capabilities, legally authorized representatives may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and Central Institutional Review Board (CIRB) regulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2030-07-29 (Estimated); Study Completion 2030-10-29 (Estimated)

PRIMARY OUTCOMES:
Major organ deterioration progression-free survival (PFS) | From date of randomization (Step 2 registration) to date of first documentation of hematologic progression, cardiac organ progression, renal organ progression, or death due to any cause, assessed up to 4 years
  Will be performed using a stratified log-rank test for comparison between study arms. The analyses will be stratified according to Mayo 2012 Prognostic Staging System for Light Chain Amyloidosis (Stage 1 versus [vs.] 2-3), hematological response following 2 cycles of daratumumab, cyclophosphamide, bortezomib and dexamethasone (Dara-VCD) induction (partial response [PR] or worse vs. very good partial response [VGPR] or better), and presence of t(11;14) by interphase fluorescence in situ hybridization [iFISH] (yes vs. no). All eligible participants will be considered in analyses of the primary endpoint, according to their assigned arm at randomization.

SECONDARY OUTCOMES:
Overall survival | From randomization to date of death due to any cause, assessed up to 4 years
  Will be performed using a stratified log-rank test for comparison between arms, with stratification according to Mayo 2012 Prognostic Staging System for Light Chain Amyloidosis (Stage 1 vs. 2-3), hematological response following 2 cycles of Dara-VCD induction (PR or worse vs. [VGPR or better), and presence of t(11;14) by iFISH (yes vs. no).
Hematologic PFS | From randomization (Step 2 registration) to date of first documentation of hematologic progression, or death due to any cause, assessed up to 4 years
  Will be performed using a stratified log-rank test for comparison between arms, with stratification according to Mayo 2012 Prognostic Staging System for Light Chain Amyloidosis (Stage 1 vs. 2-3), hematological response following 2 cycles of Dara-VCD induction (PR or worse vs. VGPR or better), and presence of t(11;14) by iFISH (yes vs. no).
Cardiac and renal organ response rates | Up to 4 years
  Progression will be defined based on objective evidence of worsening of organ dysfunction due to AL amyloid. Will be evaluated with a Cochran-Mantel-Haenszel test accounting for stratification according to Prognostic Staging System for Light Chain Amyloidosis (Stage 1 vs. 2-3), hematological response following 2 cycles of Dara-VCD induction (PR or worse vs. VGPR or better), and presence of t(11;14) by iFISH (yes vs. no).
Measurable residual disease (MRD) negativity rate | From baseline to off treatment follow-up (prior to progression) or 12 months post consolidation
  Will be evaluated with a Cochran-Mantel-Haenszel test accounting for stratification according to Prognostic Staging System for Light Chain Amyloidosis (Stage 1 vs. 2-3), hematological response following 2 cycles of Dara-VCD induction (PR or worse vs. VGPR or better), and presence of t(11;14) by iFISH (yes vs. no).
Best overall hematologic response | From date of initial registration (Step 1) and date of randomization (Step 2 registration) to date of first documentation of hematologic PR, VGPR, or CR, assessed up to 4 years
  Will be evaluated with a Cochran-Mantel-Haenszel test accounting for stratification according to Prognostic Staging System for Light Chain Amyloidosis (Stage 1 vs. 2-3), hematological response following 2 cycles of Dara-VCD induction (PR or worse vs. VGPR or better), and presence of t(11;14) by iFISH (yes vs. no).
Overall hematologic response rate | From date of initial registration (Step 1) and date of randomization (Step 2 registration) to date of first documentation of hematologic PR, VGPR, or CR, assessed up to 4 years
  Will be evaluated with a Cochran-Mantel-Haenszel test accounting for stratification according to Prognostic Staging System for Light Chain Amyloidosis (Stage 1 vs. 2-3), hematological response following 2 cycles of Dara-VCD induction (PR or worse vs. VGPR or better), and presence of t(11;14) by iFISH (yes vs. no).
Rate of complete response | Up to 4 years
  Will be evaluated with a Cochran-Mantel-Haenszel test accounting for stratification according to Prognostic Staging System for Light Chain Amyloidosis (Stage 1 vs. 2-3), hematological response following 2 cycles of Dara-VCD induction (PR or worse vs. VGPR or better), and presence of t(11;14) by iFISH (yes vs. no).
Rate of very good complete response or better | Up to 4 years
  Will be evaluated with a Cochran-Mantel-Haenszel test accounting for stratification according to Prognostic Staging System for Light Chain Amyloidosis (Stage 1 vs. 2-3), hematological response following 2 cycles of Dara-VCD induction (PR or worse vs. VGPR or better), and presence of t(11;14) by iFISH (yes vs. no).
Time to next treatment | From date of initial registration (Step 1) to date of initiation of next line of therapy, assessed up to 4 years
  Will be analyzed using the cumulative incidence competing risks method.
Change in patient reported health quality of life (QOL) | From baseline to post-maintenance, approximately 24 months
  Will use the PROMIS-29+2 (version 2.1) to compare the physical function between participants in the ASCT vs. non-ASCT arm.
Incidence of adverse events | Up to the end of maintenance therapy, approximately 24 months
  Participant-reported toxicity will be examined using Patient Reported Outcome-Common Terminology Criteria for Adverse Events.

OTHER OUTCOMES:
Bone marrow Next Generation Flow based MRD negativity rates | At the end of consolidation, approximately 6 months
  Comparisons of MRD negativity rates between arms will be made using a stratified Cochran-Mantel-Haenszel test, with analyses stratified according to European modification of the Mayo Prognostic Staging System for Light Chain Amyloidosis (Stage 1 vs. 2-3a), hematological response following 2 cycles of Dara-VCD induction (PR or worse vs. VGPR or better), and presence of t(11;14) by iFISH (yes vs. no).
Change in physical function as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS)-29+2 physical function domain | From baseline to post-consolidation, approximately 6 months
  Analysis will be conducted using multiple linear regression analysis, adjusting for the clinical study-specified stratification factors (which are also anticipated to influence QOL endpoints), and the baseline score as covariates.
Change in PROMIS-29 fatigue domain score | From baseline to post-consolidation, approximately 6 months
  Analysis will be conducted using linear regression, adjusting for the clinical study-specified stratification factors and the baseline PROMIS-29 fatigue domain score as covariates. Additionally, will conduct longitudinal modeling of the physical function domain score over time (through 12 months from registration Step 3). For longitudinal modeling, linear mixed models will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick A Hagen, Principal Investigator — SWOG Cancer Research Network
Locations (35):
- United States (35):
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Mission Cancer and Blood - Ankeny, Ankeny, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mission Cancer and Blood - Des Moines, Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin